CLINICAL TRIAL: NCT01058707
Title: A Phase I, Open Label, Dose Escalation Study of Oral Administration of Single Agent INK128 in Subjects With Advanced Malignancies Followed by an Expansion in Subjects With Measurable Disease
Brief Title: Dose Escalation Study of MLN0128 in Participants With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INK128-001; 2009-017284-42 (EudraCT Number); U1111-1187-4258 (Other: World Health Organization)
Record Dates: First submitted 2010-01-27; First posted 2010-01-29 (Estimated); Results first posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Advanced Solid Malignancies
Keywords: Solid tumors, MLN0128, TORC1/2 inhibitors
MeSH Terms: interventions — sapanisertib

STUDY DESIGN:
Intervention Model Description: The Escalation Phase was sequential and the Expansion Phase was parallel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- MLN0128 QD (Experimental): MLN0128 2 mg, 4 mg, 6 mg or 7 mg, capsule, orally, once daily (QD) in 28-day cycle in the Dose Escalation Phase until Maximum Tolerated Dose (MTD) was established (Up to 52.1 weeks).
  Interventions: Drug: MLN0128
- MLN0128 QW (Experimental): MLN0128 7 mg, 10 mg, 15 mg, 20 mg, 30 mg or 40 mg capsule, orally, once weekly (QW) in 28-day cycle in the Dose Escalation Phase until Maximum Tolerated Dose (MTD) was established (Up to 139.4 weeks).
  Interventions: Drug: MLN0128
- MLN0128 QDx3d QW (Experimental): MLN0128 6 mg, 9 mg, 12 mg, 16 mg or 20 mg capsule, orally, once daily every 3 days a week (QDx3d QW) in 28-day cycle in the Dose Escalation Phase until Maximum Tolerated Dose (MTD) was established (Up to 129.4 weeks).
  Interventions: Drug: MLN0128
- MLN0128 QDx5d QW (Experimental): MLN0128 7 mg, 10 mg or 13 mg capsule, orally, once daily every 5 days a week (QDx5d QW) in 28-day cycle in the Dose Escalation Phase until Maximum Tolerated Dose (MTD) was established (Up to 161.9 weeks).
  Interventions: Drug: MLN0128
- MLN0128 5 mg QD (Experimental): MLN0128 5 mg, capsule, orally, QD in 28-day cycle until disease progression or unacceptable toxicity in the Dose Expansion Phase (Up to 98.3 weeks).
  Interventions: Drug: MLN0128
- MLN0128 30 mg QW (Experimental): MLN0128 30 mg, capsule, orally QW in 28-day cycle until disease progression or unacceptable toxicity in the Dose Expansion Phase (Up to 240 weeks).
  Interventions: Drug: MLN0128
- MLN0128 40 mg QW (Experimental): MLN0128 40 mg, capsule, orally, QW in 28-day cycle until disease progression or unacceptable toxicity in the Dose Expansion Phase (Up to 100.1 weeks).
  Interventions: Drug: MLN0128

INTERVENTIONS:
Drug: MLN0128 — MLN0128 capsules
  Other Names: INK128; TAK-128

SUMMARY:
This is a Phase I, open label, Dose Escalation study of oral administration of single agent MLN0128 in participants with Advanced Malignancies followed by an Expansion Phase in participants with renal cell carcinoma, endometrial cancer or urothelial cancer who have measurable disease.

DETAILED DESCRIPTION:
The drug being tested in this study is called MLN0128. MLN0128 is being tested to treat people who have Advanced Malignancies.

The study enrolled approximately 198 patients. Participants were assigned to one of the following dose regimens in the Dose Escalation Phase to establish the Maximum Tolerated Dose (MTD):

* MLN0128 QD
* MLN0128 QW
* MLN0128 QDx3dQW
* MLN0128 QDx5dQW

MLN0128 capsule, orally, once daily (QD) or Once weekly (QW) in the Dose Escalation Phase until MTD was established.

Once MTD was determined, participants were then enrolled in the Dose Expansion Phase to receive:

* MLN0128 5 mg QD
* MLN0128 30 mg QW
* MLN0128 40 mg QW

This multi-centre trial was conducted worldwide. The overall time to participate in this study was approximately 244 weeks. Participants will make multiple visits to the clinic, and were contacted by telephone OR plus a final visit after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written consent
* Locally advanced or metastatic solid tumors with the exception of primary brain tumor, and have failed standard of care therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Ability to swallow oral medications
* For women of child-bearing potential, negative serum or urine pregnancy test within 14 days prior to the first study drug administration and use of physician-approved method of birth control from 30 days prior to 90 days following the last study drug administration
* Male participants must be surgically sterile or must agree to use physician-approved contraception during the study and for 90 days following the last study drug administration
* Clinical laboratory values as specified in the protocol

Additionally, to be eligible for the Dose Expansion portion of the study:

* Participants must have evidence of measurable disease per response evaluation criteria in solid tumors (RECIST) version 1.1 by radiographic techniques or magnetic resonance imaging
* Participants must have a pathologic diagnosis of advanced or recurrent endometrial adenocarcinoma and must have failed at least 1 prior line of standard chemotherapy
* Participants must have a pathologic diagnosis of advanced/metastatic urothelial cancer (carcinoma of the bladder, ureter, and/or renal pelvis) and must have failed at least 1 line of prior therapy in the metastatic/unresectable setting
* Participants must have a pathologic diagnosis of advanced renal cell carcinoma (RCC), with histological or cytological confirmation of RCC and must have failed at least 1 prior line of anti-vascular endothelial growth factor therapy (VEGF) therapy (including but not limited to sunitinib, and/or sorafenib, and/or bevacizumab and/or pazopanib, and/or axitinib) and must not have received prior therapy with a target of rapamycin complex 1 (TORC1) inhibitor (such as temsirolimus or everolimus); or
* Participants must have a pathologic diagnosis of advanced renal cell carcinoma (RCC) and must have progressed on treatment with a TORC1 inhibitor (such as temsirolimus or everolimus).

Exclusion Criteria:

* Diagnosis of primary brain tumor
* Have received prior cancer or other investigational therapy within 2 weeks prior to the first administration of study drug
* Known impaired cardiac function or clinically significant cardiac disease
* Known treatment with systemic corticosteroid within one week prior to the first administration of study drug
* Diabetes mellitus
* Human immunodeficiency virus (HIV) infection
* Known active cardiovascular disease condition as specified in protocol
* Failed to recover from the reversible effects of prior anticancer therapies
* Pregnancy (positive serum or urine pregnancy test) or breast feeding
* Malabsorption due to prior gastrointestinal (GI) surgery, GI disease
* Other clinically significant co-morbidities

Please note that there are additional inclusion and exclusion criteria. The study center will determine if you meet all of the criteria.

Site personnel will explain the trial in detail and answer any question you may have if you do qualify for the study. You can then decide whether or not you wish to participate. If you do not qualify for the trial, site personnel will explain the reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2010-01-04 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (16):
- United States (14):
  - Scottsdale, Arizona
  - Los Angeles, California
  - Miami, Florida
  - Sarasota, Florida
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Buffalo, New York
  - New York, New York
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
- Spain (2):
  - Barcelona
  - Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Voss MH, Gordon MS, Mita M, Rini B, Makker V, Macarulla T, Smith DC, Cervantes A, Puzanov I, Pili R, Wang D, Jalal S, Pant S, Patel MR, Neuwirth RL, Enke A, Shou Y, Sedarati F, Faller DV, Burris HA 3rd. Phase 1 study of mTORC1/2 inhibitor sapanisertib (TAK-228) in advanced solid tumours, with an expansion phase in renal, endometrial or bladder cancer. Br J Cancer. 2020 Nov;123(11):1590-1598. doi: 10.1038/s41416-020-01041-x. Epub 2020 Sep 11. PMID 32913286

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 15 investigative sites in Spain and the United States from 4 January 2010 to 7 February 2019.
Pre-assignment Details: Participants with a diagnosis of advanced malignancies were enrolled and received rising doses of MLN0128 in the Dose Escalation Phase to determine Maximum Tolerated Dose (MTD). In the Dose Expansion Phase participants were enrolled to receive one of 3 dose regimens: MLN0128 5 mg once daily (QD), 30 mg once weekly (QW) or 40 mg QW.
Period: Overall Study
Arm/Group | MLN0128 QD | MLN0128 QW | MLN0128 QDx3d QW | MLN0128 QDx5d QW | MLN0128 5 mg QD | MLN0128 30 mg QW | MLN0128 40 mg QW
Started | 31 | 30 | 33 | 22 | 39 | 17 | 26
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 31 | 30 | 33 | 22 | 39 | 17 | 26
Not completed — Disease Progression | 15 | 20 | 20 | 15 | 23 | 10 | 12
Not completed — Adverse Event | 11 | 4 | 7 | 6 | 7 | 3 | 1
Not completed — Subject Decision | 5 | 3 | 3 | 1 | 2 | 3 | 6
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Reason Not Specified | 0 | 3 | 2 | 0 | 7 | 1 | 7

BASELINE CHARACTERISTICS:
Population: All Participants as Treated (ASaT) population included all participants who received at least 1 dose of MLN0128.
Groups:
- Total: Total of all reporting groups
Arm/Group | MLN0128 QD | MLN0128 QW | MLN0128 QDx3d QW | MLN0128 QDx5d QW | MLN0128 5 mg QD | MLN0128 30 mg QW | MLN0128 40 mg QW | Total
Number analyzed (Participants) | 31 | 30 | 33 | 22 | 39 | 17 | 26 | 198
Age, Continuous [Mean (Full Range); unit: years] | 59.7 [24 to 75] | 53.8 [34 to 89] | 56.1 [36 to 87] | 58.1 [32 to 75] | 58.8 [30 to 81] | 59.7 [32 to 76] | 63.2 [44 to 80] | 58.31 [24 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 22 | 13 | 16 | 6 | 14 | 105
  Male | 15 | 12 | 11 | 9 | 23 | 11 | 12 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 7 | 9 | 8 | 1 | 2 | 49
  Not Hispanic or Latino | 20 | 19 | 26 | 13 | 30 | 16 | 24 | 148
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 6
  White | 28 | 29 | 30 | 22 | 37 | 17 | 25 | 188
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 18 | 19 | 12 | 32 | 15 | 25 | 142
  Spain | 10 | 12 | 14 | 10 | 7 | 2 | 1 | 56

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Phase: Maximum Tolerated Dose (MTD)
Description: MTD was defined as the highest dose level of MLN0128 at which no more than 1 out of 6 evaluable participants experienced a DLT during the first cycle (28 days) of therapy.
Time Frame: Cycle 1 (28 Days)
Population: Dose Escalation-Evaluable Population included participants who received ≥ 75% or more of planned doses of MLN0128 in Cycle 1 or stopped study drug before receiving 75% of doses because of study drug-related AEs considered a DLT.
Measure: Number; unit: milligrams (mg)
Arm/Group | MLN0128 QD | MLN0128 QW | MLN0128 QDx3d QW | MLN0128 QDx5d QW
Number analyzed (Participants) | 25 | 27 | 29 | 22
milligrams (mg) | 6 | 40 | 9 | 7

2. Primary Outcome: Dose Escalation Phase: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs were defined as MLN0128-related treatment-emergent adverse events (TEAEs) that occurred within the Cycle 1 (first 28 days of treatment) as per Common Terminology Criteria for Adverse Events (CTCAE): Any ≥Grade 3 or non-hematologic toxicity except for Grade 3 nausea and/or vomiting and diarrhea, Grade 3 hyperglycemia lasting ≤ 14 days, Grade 3 rash lasting ≤ 3 days; Grade 4 neutropenia lasting >7 days in the absence of growth factor support; Grade 4 neutropenia of any duration associated with fever ≥38.5 degree celsius and/or systemic infection; Any other Grade 4 hematologic toxicity; Inability to administer at least 75% of planned doses of MLN0128 within Cycle 1 due to drug-related toxicity and any clinically significant occurrence that the investigators and sponsor agreed would place participants at an undue safety risk.
Time Frame: Cycle 1 (28 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MLN0128 QD | MLN0128 QW | MLN0128 QDx3d QW | MLN0128 QDx5d QW
Number analyzed (Participants) | 25 | 27 | 29 | 22
Participants | 7 | 2 | 6 | 7

3. Primary Outcome: Number of Participants Experiencing One or More Treatment-Emergent Adverse Events (AEs), Serious Adverse Events (SAEs), AEs Resulting in Discontinuation of MLN0128 and Fatal AEs Within 30 Days of Last Dose of Study Drug
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. A serious adverse event is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: First dose of study drug through 30 days after the administration of the last dose of study drug (Up to approximately 244 weeks)
Population: ASaT population included all participants who received at least 1 dose of MLN0128.
Measure: Count of Participants; unit: Participants
Arm/Group | MLN0128 QD | MLN0128 QW | MLN0128 QDx3d QW | MLN0128 QDx5d QW | MLN0128 5 mg QD | MLN0128 30 mg QW | MLN0128 40 mg QW
Number analyzed (Participants) | 31 | 30 | 33 | 22 | 39 | 17 | 26
Participants
  TEAE | 31 | 30 | 33 | 22 | 39 | 17 | 26
  SAE | 13 | 10 | 17 | 10 | 19 | 6 | 9
  AEs Resulting in Discontinuation of MLN0128 | 11 | 4 | 7 | 6 | 7 | 3 | 2
  Fatal AEs within 30 Days of Last Dose Study Drug | 1 | 1 | 2 | 0 | 0 | 2 | 1

4. Primary Outcome: Dose Expansion: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieved complete response (CR) or partial response (PR based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. CR is defined as disappearance of all target lesions and PR was defined of at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD and for non-target lesions. Data was categorized as per type of cancer.
Time Frame: From the first dose of study drug up to disease progression or death (Up to approximately 240 weeks)
Population: Response-Evaluable Population included participants who received at least 1 dose of MLN0128, had measurable disease at Baseline, and underwent at least 1 post-Baseline disease assessment. Participants without a post-Baseline disease assessment but discontinued study drug due to symptomatic and/or clinical deterioration were included.
Measure: Number; unit: percentage of participants
Arm/Group | MLN0128 5 mg QD | MLN0128 30 mg QW | MLN0128 40 mg QW
Number analyzed (Participants) | 36 | 14 | 22
percentage of participants
  Cancer Type: Renal: number analyzed (Participants) | 20 | 8 | 13
  Cancer Type: Renal | 15 | 13 | 15
  Cancer Type: Endometrial: number analyzed (Participants) | 11 | 4 | 3
  Cancer Type: Endometrial | 9 | 0 | 0
  Cancer Type: Bladder: number analyzed (Participants) | 5 | 2 | 6
  Cancer Type: Bladder | 0 | 0 | 0

5. Primary Outcome: Dose Expansion Phase: Duration of Objective Response
Description: Duration of objective response is defined as the number of months from the start date of CR or PR (whichever occurred first) based on RECIST Criteria version 1.1 to the first date of objectively documented progressive disease (PD) for participants who achieved CR or PR. PD is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: From the first dose of study drug up to disease progression or death (Up to approximately 240 weeks)
Population: Response-Evaluable Population:participants who received ≥1 dose of MLN0128,had measurable disease at Baseline,had ≥1 post-Baseline disease assessment.Participants without post-Baseline disease assessment but discontinued study drug due to symptomatic and/or clinical deterioration were included.CR/PR participants with available data were analyzed.
Measure: Median (Full Range); unit: months
Arm/Group | MLN0128 5 mg QD | MLN0128 30 mg QW | MLN0128 40 mg QW
Number analyzed (Participants) | 4 | 1 | 2
months | 8.90 [3.48 to 23.06] | 56.05 [56.05 to 56.05] | 20.73 [20.24 to 21.22]

6. Primary Outcome: Dose Expansion: Duration of Stable Disease (SD)
Description: Duration of SD was evaluated for participants with best response of SD and is defined as number of months from date of first dose to date of PD. As per RECIST 1.1, SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PR was defined of at least a 30% decrease in sum of longest diameter (LD) of target lesions, taking as reference the baseline sum LD and for non-target lesions. PD is defined as at least a 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study (this includes baseline sum if that is smallest on study).
Time Frame: From the first dose of study drug up to disease progression or death (Up to approximately 240 weeks)
Population: Response-Evaluable Population: participants who received ≥1 dose of MLN0128, had measurable disease at Baseline (BL), underwent ≥1 post-BL disease assessment. Participants without post-BL disease assessment but discontinued study drug due to symptomatic and/or clinical deterioration were included. SD participants with available data were analyzed.
Measure: Median (Full Range); unit: months
Arm/Group | MLN0128 5 mg QD | MLN0128 30 mg QW | MLN0128 40 mg QW
Number analyzed (Participants) | 19 | 5 | 11
months | 3.68 [0.95 to 14.88] | 2.20 [0.76 to 5.45] | 3.55 [1.18 to 13.08]

7. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for MLN0128
Time Frame: Pre-dose and multiple time-points up to 8 hours post-dose on Day 1 of Cycles 1 and 2
Population: Pharmacokinetic (PK) population consisted of all participants included during the dose escalation phase of the study who received at least 1 dose of MLN0128. Number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Full Range); unit: ng/mL
Groups:
- MLN0128 2 mg QD: MLN0128 2 mg capsule, orally, QD in 28-day cycle (Up to 10.1 weeks).
- MLN0128 4 mg QD: MLN0128 4 mg capsule, orally, QD in 28-day cycle (Up to 14.0 weeks)
- MLN0128 6 mg QD: MLN0128 6 mg capsule, orally, QD in 28-day cycle (Up to 32.0 weeks).
- MLN0128 7 mg QD: MLN0128 7 mg, capsule, orally QD in 28-day cycle (Up to 52.1 weeks).
- MLN0128 7 mg QW: MLN0128 7 mg, capsule, orally QD in 28-day cycle (Up to 7.0 weeks).
- MLN0128 10 mg QW: MLN0128 10 mg, capsule, orally QW in 28-day cycle (Up to 15.1 weeks).
- MLN0128 15 mg QW: MLN0128 15 mg, capsule, orally QW in 28-day cycle (Up to 7.1 weeks).
- MLN0128 20 mg QW: MLN0128 20 mg, capsule, orally QW in 28-day cycle (Up to 10.1 weeks).
- MLN0128 6 mg QDx3dQW: MLN0128 6 mg, capsule, orally QDx3d QW in 28-day cycle (Up to 8.4 weeks).
- MLN0128 9 mg QDx3d QW: MLN0128 9 mg, capsule, orally QDx3d QW in 28-day cycle (Up to 129.4 weeks).
- MLN0128 12 mg QDx3d QW: MLN0128 12 mg, capsule, orally QDx3d QW in 28-day cycle (Up to 11.4 weeks).
- MLN0128 16 mg QDx3d QW: MLN0128 16 mg, capsule, orally QDx3d QW in 28-day cycle (Up to 31.4 weeks).
- MLN0128 20 mg QDx3dQW: MLN0128 20 mg, capsule, orally QDx3d QW in 28-day cycle (Up to 7.4 weeks).
- MLN0128 7 mg QDx5dQW: MLN0128 7 mg, capsule, orally QDx5d QW in 28-day cycle (Up to 15.9 weeks).
- MLN0128 10 mg QDx5dQW: MLN0128 10 mg, capsule, orally QDx5d QW in 28-day cycle (Up to 161.9 weeks).
- MLN0128 13 mg QDx5dQW: MLN0128 13 mg, capsule, orally QDx5d QW in 28-day cycle (Up to 7.7 weeks).
Arm/Group | MLN0128 2 mg QD | MLN0128 4 mg QD | MLN0128 6 mg QD | MLN0128 7 mg QD | MLN0128 7 mg QW | MLN0128 10 mg QW | MLN0128 15 mg QW | MLN0128 20 mg QW | MLN0128 30 mg QW | MLN0128 40 mg QW | MLN0128 6 mg QDx3dQW | MLN0128 9 mg QDx3d QW | MLN0128 12 mg QDx3d QW | MLN0128 16 mg QDx3d QW | MLN0128 20 mg QDx3dQW | MLN0128 7 mg QDx5dQW | MLN0128 10 mg QDx5dQW | MLN0128 13 mg QDx5dQW
Number analyzed (Participants) | 3 | 7 | 12 | 8 | 3 | 3 | 3 | 3 | 3 | 15 | 3 | 8 | 6 | 11 | 4 | 6 | 11 | 3
ng/mL
  Cycle 1 Day 1 | 13.7 [12.30 to 16.30] | 20.5 [9.54 to 35.70] | 48.9 [18.60 to 75.60] | 67.8 [21.10 to 143.00] | 43.6 [16.20 to 94.40] | 75.9 [43.60 to 139.00] | 80.2 [24.30 to 173.00] | 136.6 [66.80 to 217.00] | 174.0 [101.00 to 259.00] | 193.8 [57.90 to 358.00] | 88.5 [72.90 to 115.00] | 82.9 [25.00 to 111.00] | 124.3 [50.90 to 320.00] | 78.5 [35.20 to 184.00] | 194.0 [118.00 to 300.00] | 46.9 [18.80 to 79.00] | 48.5 [22.60 to 76.50] | 110.1 [42.30 to 181.00]
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 5 | 7 | 3 | 2 | 2 | 3 | 1 | 3 | 8 | 3 | 5 | 3 | 9 | 1 | 4 | 7 | 1
  Cycle 2 Day 1 | 16.2 [12.00 to 22.70] | 22.1 [11.90 to 35.90] | 39.4 [24.00 to 76.40] | 65.0 [28.20 to 130.00] | 66.7 [55.80 to 77.60] | 40.5 [22.40 to 58.50] | 66.9 [47.70 to 87.90] | 134.00 [134.00 to 134.00] | 142.6 [96.70 to 222.00] | 249.8 [140.00 to 394.00] | 60.0 [52.50 to 74.40] | 87.7 [46.80 to 118.00] | 115.1 [93.40 to 143.00] | 113.6 [42.50 to 292.00] | 183.00 [183.00 to 183.00] | 60.1 [23.50 to 126.00] | 60.0 [32.00 to 95.70] | 96.50 [96.50 to 96.50]

8. Secondary Outcome: Ctrough: Observed Concentration at the End of a Dosing Interval
Time Frame: Pre-dose and multiple time-points up to 8 hours post-dose on Day 1 of Cycles 1 and 2
Population: PK population consisted of all participants included during the dose escalation phase of the study who received at least 1 dose of MLN0128. Number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | MLN0128 2 mg QD | MLN0128 4 mg QD | MLN0128 6 mg QD | MLN0128 7 mg QD | MLN0128 7 mg QW | MLN0128 10 mg QW | MLN0128 15 mg QW | MLN0128 20 mg QW | MLN0128 30 mg QW | MLN0128 40 mg QW | MLN0128 6 mg QDx3dQW | MLN0128 9 mg QDx3d QW | MLN0128 12 mg QDx3d QW | MLN0128 16 mg QDx3d QW | MLN0128 20 mg QDx3dQW | MLN0128 7 mg QDx5dQW | MLN0128 10 mg QDx5dQW | MLN0128 13 mg QDx5dQW
Number analyzed (Participants) | 3 | 7 | 12 | 8 | 3 | 3 | 3 | 3 | 3 | 15 | 3 | 8 | 6 | 11 | 4 | 6 | 11 | 3
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 7 | 11 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 8 | 6 | 11 | 4 | 6 | 9 | 3
  Cycle 1 Day 1 | 0.9 [0.00 to 2.76] | 1.2 [0.00 to 2.48] | 3.5 [0.00 to 8.84] | 4.4 [1.15 to 9.22] |  |  |  |  |  |  | 2.5 [0.00 to 5.01] | 6.8 [0.00 to 16.80] | 9.9 [1.83 to 22.90] | 8.1 [0.00 to 21.50] | 44.7 [6.35 to 123.00] | 3.1 [2.02 to 4.48] | 3.6 [0.00 to 10.10] | 21.7 [5.85 to 43.70]
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 5 | 7 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 2 | 9 | 1 | 4 | 6 | 1
  Cycle 2 Day 1 | 4.5 [1.48 to 9.76] | 3.7 [0.00 to 10.30] | 4.5 [3.07 to 9.37] | 3.0 [1.24 to 6.23] |  |  |  |  |  |  | 10.3 [0.00 to 25.10] | 10.8 [5.03 to 25.50] | 4.4 [3.34 to 5.38] | 10.0 [0.00 to 27.10] | 11.40 [11.40 to 11.40] | 5.2 [1.82 to 11.20] | 3.0 [1.08 to 4.68] | 6.58 [6.58 to 6.58]

9. Secondary Outcome: Terminal Phase Elimination Half-life (T1/2) for MLN0128
Time Frame: Pre-dose and multiple time-points up to 8 hours post-dose on Day 1 of Cycles 1 and 2
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | MLN0128 2 mg QD | MLN0128 4 mg QD | MLN0128 6 mg QD | MLN0128 7 mg QD | MLN0128 7 mg QW | MLN0128 10 mg QW | MLN0128 15 mg QW | MLN0128 20 mg QW | MLN0128 30 mg QW | MLN0128 40 mg QW | MLN0128 6 mg QDx3dQW | MLN0128 9 mg QDx3d QW | MLN0128 12 mg QDx3d QW | MLN0128 16 mg QDx3d QW | MLN0128 20 mg QDx3dQW | MLN0128 7 mg QDx5dQW | MLN0128 10 mg QDx5dQW | MLN0128 13 mg QDx5dQW
Number analyzed (Participants) | 3 | 7 | 12 | 8 | 3 | 3 | 3 | 3 | 3 | 15 | 3 | 8 | 6 | 11 | 4 | 6 | 11 | 3
hours
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 4 | 10 | 4 | 1 | 2 | 2 | 3 | 3 | 14 | 2 | 5 | 6 | 8 | 2 | 6 | 8 | 2
  Cycle 1 Day 1 | 10.3 [10.30 to 10.30] | 7.4 [5.27 to 8.22] | 6.3 [4.86 to 10.40] | 6.2 [5.66 to 6.23] | 6.47 [6.47 to 6.47] | 5.8 [5.72 to 5.95] | 9.4 [6.99 to 11.90] | 5.7 [4.11 to 11.60] | 5.5 [5.30 to 6.94] | 7.1 [4.07 to 12.70] | 5.5 [5.15 to 5.93] | 7.9 [6.53 to 8.12] | 6.4 [4.71 to 11.10] | 7.2 [4.59 to 9.52] | 5.5 [5.10 to 5.84] | 7.8 [5.26 to 9.38] | 6.5 [4.72 to 10.10] | 8.7 [8.20 to 9.16]
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 3 | 6 | 3 | 2 | 0 | 1 | 1 | 2 | 5 | 2 | 4 | 2 | 7 | 1 | 3 | 6 | 1
  Cycle 2 Day 1 | 8.1 [7.49 to 8.75] | 9.7 [9.47 to 11.70] | 7.9 [5.83 to 8.06] | 4.9 [3.99 to 7.85] | 5.6 [4.91 to 6.19] |  | 8.01 [8.01 to 8.01] | 4.57 [4.57 to 4.57] | 5.7 [5.08 to 6.35] | 5.6 [4.29 to 9.02] | 9.1 [6.05 to 12.10] | 7.0 [6.01 to 7.85] | 4.9 [4.63 to 5.11] | 6.4 [3.61 to 10.30] | 6.28 [6.28 to 6.28] | 6.8 [6.18 to 7.14] | 5.6 [4.19 to 7.58] | 6.42 [6.42 to 6.42]

10. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for MLN0128
Time Frame: Pre-dose and multiple time-points up to 8 hours post-dose on Day 1 of Cycles 1 and 2
Population: as for outcome 8
Measure: Mean (Full Range); unit: ng*hr/mL
Arm/Group | MLN0128 2 mg QD | MLN0128 4 mg QD | MLN0128 6 mg QD | MLN0128 7 mg QD | MLN0128 7 mg QW | MLN0128 10 mg QW | MLN0128 15 mg QW | MLN0128 20 mg QW | MLN0128 30 mg QW | MLN0128 40 mg QW | MLN0128 6 mg QDx3dQW | MLN0128 9 mg QDx3d QW | MLN0128 12 mg QDx3d QW | MLN0128 16 mg QDx3d QW | MLN0128 20 mg QDx3dQW | MLN0128 7 mg QDx5dQW | MLN0128 10 mg QDx5dQW | MLN0128 13 mg QDx5dQW
Number analyzed (Participants) | 3 | 7 | 12 | 8 | 3 | 3 | 3 | 3 | 3 | 15 | 3 | 8 | 6 | 11 | 4 | 6 | 11 | 3
ng*hr/mL
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 4 | 10 | 4 | 1 | 2 | 2 | 3 | 3 | 14 | 2 | 5 | 6 | 8 | 2 | 6 | 8 | 2
  Cycle 1 Day 1 | 185.00 [185.00 to 185.00] | 205.3 [145.00 to 269.00] | 390.6 [263.00 to 608.00] | 459.5 [195.00 to 585.00] | 440.00 [440.00 to 440.00] | 609.0 [241.00 to 977.00] | 1014.5 [179.00 to 1850.00] | 1172.7 [563.00 to 2190.00] | 1316.3 [759.00 to 2290.00] | 2149.8 [844.00 to 4310.00] | 494.0 [411.00 to 577.00] | 725.2 [388.00 to 903.00] | 922.8 [383.00 to 1470.00] | 820.1 [389.00 to 1220.00] | 1245.0 [1080.00 to 1410.00] | 326.2 [240.00 to 423.00] | 388.5 [231.00 to 761.00] | 941.5 [483.00 to 1400.00]
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1 |  |  |  |  | 371.0 [354.00 to 388.00] |  | 510.00 [510.00 to 510.00] | 1030.00 [1030.00 to 1030.00] | 1427.5 [745.00 to 2110.00] | 2876.6 [903.00 to 6110.00] |  |  |  |  |  |  |  |

11. Secondary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for MLN0128
Time Frame: Pre-dose and multiple time-points up to 8 hours post-dose on Day 1 of Cycles 1 and 2
Population: as for outcome 8
Measure: Mean (Full Range); unit: ng*hr/mL
Arm/Group | MLN0128 2 mg QD | MLN0128 4 mg QD | MLN0128 6 mg QD | MLN0128 7 mg QD | MLN0128 7 mg QW | MLN0128 10 mg QW | MLN0128 15 mg QW | MLN0128 20 mg QW | MLN0128 30 mg QW | MLN0128 40 mg QW | MLN0128 6 mg QDx3dQW | MLN0128 9 mg QDx3d QW | MLN0128 12 mg QDx3d QW | MLN0128 16 mg QDx3d QW | MLN0128 20 mg QDx3dQW | MLN0128 7 mg QDx5dQW | MLN0128 10 mg QDx5dQW | MLN0128 13 mg QDx5dQW
Number analyzed (Participants) | 3 | 7 | 12 | 8 | 3 | 3 | 3 | 3 | 3 | 15 | 3 | 8 | 6 | 11 | 4 | 6 | 11 | 3
ng*hr/mL
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 3 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 1 | 0
  Cycle 1 Day 1 | 65.4 [64.00 to 66.80] | 65.3 [51.60 to 89.80] | 95.30 [95.30 to 95.30] |  | 72.80 [72.80 to 72.80] | 106.00 [106.00 to 106.00] |  |  |  |  | 162.00 [162.00 to 162.00] | 207.5 [198.00 to 217.00] |  | 130.2 [93.40 to 167.00] |  |  | 221.00 [221.00 to 221.00] |
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Cycle 2 Day 1 |  | 62.2 [56.30 to 68.00] |  |  |  | 105.00 [105.00 to 105.00] |  |  |  |  | 182.00 [182.00 to 182.00] |  |  | 197.00 [197.00 to 197.00] |  |  |  |

12. Secondary Outcome: Tmax: Time to Maximum Observed Plasma Concentration for MLN0128
Time Frame: Pre-dose and multiple time-points up to 8 hours post-dose on Day 1 of Cycles 1 and 2
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Groups:
- MLN0128 30mg QW: MLN0128 30 mg, capsule, orally QW in 28-day cycle (Up to 139.4 weeks).
Arm/Group | MLN0128 2 mg QD | MLN0128 4 mg QD | MLN0128 6 mg QD | MLN0128 7 mg QD | MLN0128 7 mg QW | MLN0128 10 mg QW | MLN0128 15 mg QW | MLN0128 20 mg QW | MLN0128 30mg QW | MLN0128 40 mg QW | MLN0128 6 mg QDx3dQW | MLN0128 9 mg QDx3d QW | MLN0128 12 mg QDx3d QW | MLN0128 16 mg QDx3d QW | MLN0128 20 mg QDx3dQW | MLN0128 7 mg QDx5dQW | MLN0128 10 mg QDx5dQW | MLN0128 13 mg QDx5dQW
Number analyzed (Participants) | 3 | 7 | 12 | 8 | 3 | 3 | 3 | 3 | 3 | 15 | 3 | 8 | 6 | 11 | 4 | 6 | 11 | 3
hours
  Cycle 1 Day 1 | 2.0 [2.00 to 2.05] | 2.0 [0.98 to 4.00] | 1.0 [0.50 to 4.17] | 1.5 [0.50 to 7.57] | 2.1 [0.52 to 8.00] | 1.0 [1.00 to 1.97] | 2.0 [1.07 to 2.00] | 2.0 [1.00 to 2.15] | 1.0 [1.00 to 4.00] | 2.4 [1.00 to 4.53] | 0.6 [0.50 to 1.15] | 1.1 [0.55 to 4.33] | 2.0 [0.55 to 4.05] | 2.1 [0.50 to 8.67] | 3.1 [0.53 to 4.05] | 1.2 [0.50 to 4.08] | 4.0 [0.53 to 4.33] | 2.1 [1.08 to 8.00]
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 5 | 7 | 3 | 2 | 2 | 3 | 1 | 3 | 8 | 3 | 5 | 3 | 9 | 1 | 4 | 7 | 1
  Cycle 2 Day 1 | 2.0 [1.97 to 2.00] | 3.8 [1.00 to 4.03] | 2.0 [1.03 to 4.42] | 4.0 [1.00 to 4.03] | 1.02 [1.02 to 1.02] | 2.9 [1.80 to 4.00] | 2.0 [2.00 to 8.00] | 4.0 [4.00 to 4.00] | 4.0 [1.03 to 7.92] | 2.0 [1.00 to 8.00] | 4.0 [1.00 to 4.00] | 2.1 [0.50 to 7.57] | 3.7 [1.00 to 4.18] | 2.1 [0.53 to 8.00] | 1.0 [1.00 to 1.00] | 1.5 [0.97 to 7.42] | 2.0 [0.52 to 3.58] | 2.02 [2.02 to 2.02]

13. Secondary Outcome: Percentage Area Under Plasma Concentration Time Curve Extrapolated
Time Frame: Pre-dose and multiple time-points up to 8 hours post-dose on Day 1 of Cycles 1 and 2
Population: The study was acquired from another organization and limited results data are available.
Arm/Group | MLN0128 2 mg QD | MLN0128 4 mg QD | MLN0128 6 mg QD | MLN0128 7 mg QD | MLN0128 7 mg QW | MLN0128 10 mg QW | MLN0128 15 mg QW | MLN0128 20 mg QW | MLN0128 30 mg QW | MLN0128 40 mg QW | MLN0128 6 mg QDx3dQW | MLN0128 9 mg QDx3d QW | MLN0128 12 mg QDx3d QW | MLN0128 16 mg QDx3d QW | MLN0128 20 mg QDx3dQW | MLN0128 7 mg QDx5dQW | MLN0128 10 mg QDx5dQW | MLN0128 13 mg QDx5dQW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Percentage Change From Baseline in Eukaryotic Initiation Factor 4E-binding Protein 1 (P4EBP1), Serine/Threonine Protein Kinase B (PAKT) and Ribosomal Protein S6 (PS6)
Description: P4EBP, PAKT and PS6 were assayed in skin biopsies. A negative percentage change from Baseline indicates improvement.
Time Frame: Baseline, Cycle 1 Week 2
Population: ASaT population included all participants who received at least 1 dose of MLN0128 in dose escalation phase. Participants with data at Baseline and Cycle 1 Week 2 are included. Number analyzed is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | MLN0128 QD | MLN0128 QW | MLN0128 QDx3d QW | MLN0128 QDx5d QW
Number analyzed (Participants) | 31 | 30 | 33 | 22
percentage change
  p4EBP1: number analyzed (Participants) | 19 | 23 | 27 | 16
  p4EBP1 | -64.1 (47.65) | -15.5 (378.88) | -99.5 (2.75) | 87.4 (43.83)
  pAKT: number analyzed (Participants) | 20 | 22 | 25 | 14
  pAKT | 27.1 (73.78) | 26.9 (139.75) | 73.3 (115.55) | 168.9 (514.88)
  pS6: number analyzed (Participants) | 21 | 24 | 27 | 16
  pS6 | -50.2 (43.89) | -42.7 (59.64) | -68.2 (37.98) | -82.5 (12.15)

ADVERSE EVENTS:
Time Frame: All cause-mortality were collected throughout the study; SAEs and Other (non-serious) were collected from the first dose of study drug plus 30 days after last dose of study drug (Up to approximately 244 weeks)
Arm/Group | MLN0128 QD | MLN0128 QW | MLN0128 QDx3d QW | MLN0128 QDx5d QW | MLN0128 5 mg QD | MLN0128 30 mg QW | MLN0128 40 mg QW
All-Cause Mortality (participants affected / at risk) | 3/31 | 2/30 | 2/33 | 0/22 | 2/39 | 2/17 | 3/26
Serious Adverse Events (participants affected / at risk) | 13/31 | 10/30 | 17/33 | 10/22 | 19/39 | 6/17 | 9/26
Other Adverse Events (participants affected / at risk) | 31/31 | 30/30 | 33/33 | 22/22 | 39/39 | 17/17 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MLN0128 QD (N=31) | MLN0128 QW (N=30) | MLN0128 QDx3d QW (N=33) | MLN0128 QDx5d QW (N=22) | MLN0128 5 mg QD (N=39) | MLN0128 30 mg QW (N=17) | MLN0128 40 mg QW (N=26)
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 4 | 2 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 3 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with MLN0128 10 mg QW escalation phase and is not related. One treatment-emergent death occurred during treatment with MLN0128 9 mg QDx3dQW escalation phase and is not related.
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with MLN0128 12 mg QDx3dQW escalation phase and is not related.
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with MLN0128 7 mg QD escalation phase and is not related.
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 1 | 0 | 2 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 — One treatment-emergent death occurred during treatment with MLN0128 30 mg QW expansion phase and is not related.
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with MLN0128 6 mg QD in escalation phase and is not related.
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with MLN0128 6 mg QD escalation phase and is related.
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with MLN0128 6 mg QD escalation phase and is related.
Renal failure (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 2
Carcinoid syndrome (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with MLN0128 40 mg QW expansion phase and is not related.
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with MLN0128 40 mg QW expansion phase and is not related.
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1 — One treatment-emergent death occurred during treatment with MLN0128 30 mg QW expansion phase and is not related. One treatment-emergent death occurred during treatment with MLN0128 40 mg QW expansion phase and is not related.
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0 | 0 — One treatment-emergent death occurred during treatment with MLN0128 5 mg QD expansion phase and is not related.
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MLN0128 QD (N=31) | MLN0128 QW (N=30) | MLN0128 QDx3d QW (N=33) | MLN0128 QDx5d QW (N=22) | MLN0128 5 mg QD (N=39) | MLN0128 30 mg QW (N=17) | MLN0128 40 mg QW (N=26)
Nausea (Gastrointestinal disorders) | 16 | 22 | 24 | 13 | 21 | 12 | 20
Vomiting (Gastrointestinal disorders) | 12 | 20 | 20 | 12 | 12 | 9 | 20
Stomatitis (Gastrointestinal disorders) | 11 | 10 | 22 | 13 | 19 | 9 | 11
Diarrhoea (Gastrointestinal disorders) | 14 | 10 | 17 | 9 | 20 | 9 | 11
Dry mouth (Gastrointestinal disorders) | 8 | 7 | 3 | 2 | 5 | 3 | 7
Abdominal pain (Gastrointestinal disorders) | 3 | 6 | 4 | 4 | 8 | 6 | 4
Constipation (Gastrointestinal disorders) | 1 | 6 | 6 | 3 | 10 | 8 | 10
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 2 | 2 | 3 | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 3 | 2 | 1 | 0 | 2 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 2 | 3 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 0 | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 2 | 0 | 5
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 26 | 18 | 22 | 12 | 18 | 12 | 20
Decreased appetite (Metabolism and nutrition disorders) | 13 | 12 | 20 | 9 | 20 | 7 | 14
Dehydration (Metabolism and nutrition disorders) | 5 | 6 | 6 | 1 | 7 | 4 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 4 | 2 | 5 | 6 | 3 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 | 1 | 4 | 2 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 3 | 4 | 3 | 4 | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2 | 4 | 1 | 3 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 1 | 2 | 2 | 3 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 1 | 1 | 2
Hypocholesterolaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 7 | 15 | 13 | 10 | 7 | 2 | 5
Fatigue (General disorders) | 10 | 9 | 15 | 7 | 25 | 11 | 24
Pyrexia (General disorders) | 2 | 9 | 8 | 6 | 8 | 1 | 5
Chills (General disorders) | 1 | 3 | 3 | 2 | 2 | 0 | 3
Oedema peripheral (General disorders) | 3 | 4 | 0 | 1 | 9 | 1 | 5
Chest pain (General disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 0
Performance status decreased (General disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 8 | 9 | 5 | 4 | 3 | 6
Dysgeusia (Nervous system disorders) | 9 | 4 | 4 | 4 | 10 | 4 | 3
Dizziness (Nervous system disorders) | 4 | 3 | 5 | 1 | 9 | 1 | 3
Tremor (Nervous system disorders) | 2 | 0 | 3 | 3 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 2 | 2 | 0 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 3 | 0 | 1 | 0 | 2 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 10 | 4 | 7 | 4 | 1 | 0 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 10 | 0 | 6 | 2 | 12 | 5 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3 | 1 | 4 | 10 | 1 | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 4 | 0 | 3 | 1 | 3 | 0 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 3 | 3 | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 2 | 17 | 4 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 1 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 13 | 3 | 1 | 5 | 2 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 3 | 5 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 2 | 2 | 2 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 0 | 2 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 1 | 4 | 1 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 0 | 1 | 1 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 2 | 1 | 3
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 4 | 3 | 6 | 6 | 6 | 2 | 8
Upper respiratory tract infection (Infections and infestations) | 1 | 5 | 1 | 2 | 0 | 1 | 3
Cellulitis (Infections and infestations) | 3 | 2 | 0 | 0 | 2 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 3 | 1 | 1 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 4 | 0 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 2 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 1 | 2
Catheter site infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 10 | 4 | 7 | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 4 | 4 | 9 | 6 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 2 | 4 | 1 | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 3 | 2 | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0 | 3 | 1 | 3
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0 | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 3 | 2 | 2
Blood creatinine increased (Investigations) | 9 | 4 | 3 | 1 | 6 | 4 | 5
Weight decreased (Investigations) | 3 | 3 | 5 | 2 | 6 | 3 | 7
Blood urea increased (Investigations) | 2 | 2 | 1 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 2 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 1 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 2 | 1 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Blood urea decreased (Investigations) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 6 | 5 | 10 | 3 | 5 | 2 | 11
Lymphopenia (Blood and lymphatic system disorders) | 5 | 4 | 3 | 2 | 3 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 1 | 1 | 1 | 3 | 1 | 2
Confusional state (Psychiatric disorders) | 5 | 1 | 3 | 2 | 4 | 0 | 3
Insomnia (Psychiatric disorders) | 3 | 1 | 3 | 3 | 2 | 3 | 5
Anxiety (Psychiatric disorders) | 2 | 2 | 4 | 1 | 3 | 3 | 3
Depression (Psychiatric disorders) | 2 | 0 | 2 | 0 | 1 | 4 | 3
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 3 | 0 | 2 | 3 | 1 | 4
Dysuria (Renal and urinary disorders) | 0 | 1 | 2 | 2 | 1 | 0 | 3
Proteinuria (Renal and urinary disorders) | 0 | 2 | 2 | 0 | 0 | 1 | 3
Hypotension (Vascular disorders) | 0 | 5 | 2 | 1 | 1 | 2 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 3
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 3
Palpitations (Cardiac disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 3
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Coeliac disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 8 | 5 | 4 | 2 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 3
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 3
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 3
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 5 | 0 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 2
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 4
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 2
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Blindness transient (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device breakage (Product Issues) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT01058707/Prot_000.pdf
  • Statistical Analysis Plan (2014-01-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT01058707/SAP_001.pdf